CLINICAL TRIAL: NCT05487222
Title: Goal Directed Fluid Therapy Compared to Liberal Fluid Therapy in Patients Subjected to Colorectal Surgery
Brief Title: Goal Directed and Liberal Fluid Therapy
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Gad mostafa, Assistant professor, Mansoura University
Other Study IDs: R.19.12.704
Record Dates: First submitted 2021-12-28; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Fluid Therapy
Keywords: fluid therapy, goal directed , liberal , colorectal surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- • Liberal fluid group (L group) using traditional technique of fluid administration
  Interventions: Device: ICON
- • Goal directed fluid group(G group) using stroke volume optimization
  Interventions: Device: ICON

INTERVENTIONS:
Device: ICON — hemodynamics variability in response to different fluid regiemens

SUMMARY:
The aim is to compare intraoperative goal directed fluid therapy (GDFT) versus liberal fluid therapy in patients undergoing elective colorectal surgery by using noninvasive electrical cardiometry. This study hypothesized that GDFT is better than liberal fluid therapy to provide sufficient intra-vascular fluid volume for adequate perfusion without impairing glycolcalyx function with fluid overload

DETAILED DESCRIPTION:
Intraoperative fluid management for major abdominal and intestinal surgeries is quite important in terms of postoperative organ perfusion and complications. Many complications such as acute renal failure, hypotension, arrhythmia, and anastomosis leak may occur secondary to intraoperative hypovolemia whereas hypervolemia may cause pulmonary edema, postoperative pneumonia, prolonged mechanical ventilation, delayed wound healing, edema in the gastrointestinal system (GIS), and decreased GIS motility.

In the perioperative period, fluid therapy and gastrointestinal function may complement each other or complicate it. If fluid therapy is not optimal, it may cause delayed gastrointestinal function and avoid early oral intake. If gastrointestinal dysfunction develops in the perioperative period, it may lead to fluid and electrolyte loss and metabolic problems. Thus, the intraoperative fluid management of the patient is very important.

Accurate assessment of a patient's volume status is an important goal for the anesthetist in the operating theatre to achieve hemodynamic stability and adequate tissue oxygenation. Different intraoperative fluid management protocols are in use for this purpose. The most common one is conventional fluid management (CFM). Fluid replacement is managed according to clinical assessment and heart rate (HR), arterial blood pressure (ABP) and central venous pressure (CVP) monitorization.

While goal-directed fluid therapy (GDFT) is a perioperative strategy, where fluid administration targets continuously-measured hemodynamic variables, such as cardiac output, stroke volume, stroke volume variation, pulse pressure variation and other factors to guide intravenous and inotropic therapy, with the aim of maximizing tissue perfusion and oxygen delivery.

Cardiac output is assessed by static indices or dynamic indices. Static indices of cardiac preload such as central venous pressure (CVP) and pulmonary artery wedge pressure are of little help for decisions regarding volume replacement. Dynamic variables such as pulse pressure variation (PPV) and stroke volume variation (SVV) are increasingly used to detect the cyclic ﬂuctuation of the arterial pressure wave in the mechanically ventilated patient in order to predict ﬂuid responsiveness.

Direct measurement of SV using noninvasive techniques has become an accepted tool for stroke volume optimization and guiding fluid administration in highly risk surgical patients. Many technologies are used to measure stroke volume, including Doppler monitoring, bio impedance/reactance measurements, and arterial waveform analysis. So, when stroke volume optimization is used as the end point, it could improve the outcomes for surgical patients with good prediction of fluid administration.

Impedance cardiography (ICG) is an accurate technique for noninvasive determination of hemodynamic variables such as stroke volume (SV), stroke volume index (SVI), cardiac output (COP), cardiac index (CI), systemic vascular resistance (SVR), and systolic time ratio (STR). ICG use electrical impedance changes to generate waveform that depend on volume and velocity of blood injected into aorta as well as the force and rate of left ventricle contraction. From that curve beside heart rate and blood pressure, stroke volume ,COP ,SVR and other hemodynamic parameter are derived

ELIGIBILITY:
Inclusion Criteria:

* • patients scheduled for elective colorectal surgery

  * with (ASA) physical status I - II - of both gender aged 18-60 years old
  * Hb >12 g/dl & Hct >38%.

Exclusion Criteria:

* • Patient refusal

  * Patients with major cardiovascular problems with ejection fraction < 40 %
  * Renal impairment with serum creatinine >1.8 mg/dl .
  * Patients with hepatic dysfunction and coagulopathy.
  * Metabolic disorder, serum lactate > 4 mmol/L.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This prospective, randomized, controlled study was conducted after a written informed consent will be obtained from all participants
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
serum creatinine level | 24 hours postoperative
  mg/dl

SECONDARY OUTCOMES:
stroke volume (SV) | Basal preoperative, before induction of anesthesia (T1), just before skin incision (T2), then every 30 min until end of surgery then every 6 hour for 24 hours
stroke volume variation (SVV) | Basal preoperative, before induction of anesthesia (T1), just before skin incision (T2), then every 30 min until end of surgery then every 6 hour for 24 hours
  percentage
stroke volume index (SVI) | Basal preoperative, before induction of anesthesia (T1), just before skin incision (T2), then every 30 min until end of surgery then every 6 hour for 24 hours
  ml/m2
cardiac index | Basal preoperative, before induction of anesthesia (T1), just before skin incision (T2), then every 30 min until end of surgery then every 6 hour for 24 hours
  L/minute/m2
cardiac output (COP) | Basal preoperative, before induction of anesthesia (T1), just before skin incision (T2), then every 30 min until end of surgery then every 6 hour for 24 hours
  L/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Oncology Center, Al Mansurah, Eldakahlia, Egypt